CLINICAL TRIAL: NCT02166866
Title: Phase I/II Cancer Caregiver Interventions to Improve Quality of Life and Prevent Burnout
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1295
Record Dates: First submitted 2014-06-06; First posted 2014-06-18 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Cancer Care Recipient
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Experimental arm
  Interventions: Other: Quality of Life Questionairre and Education

INTERVENTIONS:
Other: Quality of Life Questionairre and Education

SUMMARY:
This study defines cancer caregivers as unpaid individuals who provide physical, practical, and/or emotional care and support to the cancer patient in the home setting. They may participate in this study if care recipients and the caregiver are both adults (18 years or older), with the patient having been diagnosed with cancer.The 8 intervention sessions will target the five domains of Quality Of Life (emotional, physical, social, cognitive, and spiritual well-being), be provided in group settings, and be delivered in two 45-minute sessions each week over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Ability to speak, read, write and understand English language
* Has cancer caregiver status defined as an unpaid individual who provides physical, practical, and/or emotional care and support to a cancer care recipient in the home or other healthcare setting.
* Has a care recipient:

  * ≥ 18 years of age who
  * has a malignancy (either solid tumor or hematologic) diagnosis.
  * who has signed a research authorization form
  * who is undergoing or in the last 6 months has undergone cancer treatment
* Ability to use and access to a computer, tablet or other device with internet access and video capabilities

Exclusion Criteria:

* Diagnosis within the past 12 months of active substance abuse (alcohol or drugs)
* Diagnosis within the past 12 months of active mental health condition that has required psychiatric hospitalization
* Diagnosis within the past 12 months of suicidal thoughts or attempt
* Care recipient is currently participating in another psychosocial clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers will be recruited through the Mayo Clinic inpatient and outpatient services, including but not limited to referrals from staff of the Divisions of Medical Oncology, Hematology, and Radiation Oncology and other clinics in the outpatient setting, and Divisions of HospitalMedicine, Hospice and Palliative Medicine, and other inpatient services in the hospital setting. This population was chosen as they are likely to experience caregiver-related distress for which the intervention will be beneficial.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2015-05-05 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
calculate the average number of caregivers participating in each offered web-based session | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Lapid MI, Atherton PJ, Kung S, Clark MM, Sloan JA, Whitford KJ, Hubbard JM, Gentry MT, Miller JJ, Rummans TA. A feasibility study of virtual group therapy to improve quality of life of cancer caregivers. J Psychosoc Oncol. 2022;40(6):854-867. doi: 10.1080/07347332.2021.2000550. Epub 2021 Nov 29. PMID 34842060